CLINICAL TRIAL: NCT00822328
Title: Effects of a Fermented Milk Drink Containing Lactobacillus Casei Strain Shirota on the Human Intestinal Microflora
Brief Title: Fermented Milk Drink on Human Intestinal Microflora
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cheng Hsin Rehabilitation Medical Center (Other)
Responsible Party: Yi-Hsien Lin, Division of Radiotherapy, Cheng Hsin Rehabilitation Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CHGH-IRB(173)97B-13-1
Record Dates: First submitted 2009-01-09; First posted 2009-01-14 (Estimated); Results first posted 2009-08-19 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-08

CONDITIONS: Signs and Symptoms, Digestive
Keywords: Probiotics; Lactobacillus; Intestine; Flora
MeSH Terms: conditions — Signs and Symptoms, Digestive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Fermented milk with Lactobacillus casei strain Shirota 100ml per day
  Interventions: Dietary Supplement: Yakult®300; Dietary Supplement: Lactobacillus casei strain Shirota
- 2 (Placebo Comparator): Unfermented milk without Lactobacillus casei strain Shirota 100ml per day
  Interventions: Dietary Supplement: Yakult®300

INTERVENTIONS:
Dietary Supplement: Yakult®300 — Yakult®300 was given 100 ml once per day for four weeks.
  Fermented or unfermented milk per 100 ml bottle per day for four week.
Dietary Supplement: Lactobacillus casei strain Shirota — Lactobacillus casei strain Shirota
  Arms: 1

SUMMARY:
Fermented milk is a popular drink. Recent studies revealed that some fermented milk containing some strains of lactic acid bacteria have health-promoting effects through improvement of the intestinal microflora and modulation of the immune system. Lactobacillus casei strain Shirota (LcS) is a probiotic bacterium used in the production of fermented milk products and lactic acid bacteria preparations. LcS has been shown to modify allergen-induced immune responses in allergic rhinitis, altering fermentation patterns in the small bowel, prevention of recurrent urinary tract infections in women. Yakult®300 is a fermented milk containing at least 3x10^10 live LcS cells per 100 ml bottle. This study aimed to evaluate the effects of a fermented milk drink containing Lactobacillus casei strain Shirota on the human intestinal microflora.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers and willing to give voluntary written informed consent

Exclusion Criteria:

* Major systemic disease
* Pregnancy, parturient and feeding woman, or expect to be pregnant
* Abnormal liver function
* Abnormal renal function
* Abnormal gastrointestinal function
* Take medication for gastrointestinal function
* Stroke, myocardial infarction,
* Poor compliance for study protocol

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hsien Lin, M.D., Principal Investigator — Division of Radiotherapy, Cheng Hsin Rehabilitation Medical Center
Locations (1):
- Division of Radiotherapy, Cheng Hsin Rehabilitation Medical Center, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 healthy volunteers were recuited on Jan.11, 2009 at Cheng Hsin Rehabilitation Medical Center.
Groups:
- Fermented Milk (Study Group): Fermented milk with Lactobacillus casei strain Shirota 100ml per day
- Unfermented Milk (Placebo Group): Unfermented milk without Lactobacillus casei strain Shirota 100ml per day
Period: Overall Study
Arm/Group | Fermented Milk (Study Group) | Unfermented Milk (Placebo Group)
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fermented Milk (Study Group) | Unfermented Milk (Placebo Group) | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.00 (3.54) | 32.42 (6.33) | 31.21 (5.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  Taiwan | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Modification of the Composition of the Intestinal Microflora: Bifidobacterium
Description: Fecal specimens were obtained from all 24 healthy volunteers at week 0, 1, 2, 3, 4, 5, 6. Bifidobacterium was cultured. Bacterial colonies were counted.
Time Frame: week 0, 1, 2, 3, 4, 5, 6.
Population: The number of participants for analysis was per protocol analysis.
Measure: Log Mean (Standard Deviation); unit: log10 CFU/g
Arm/Group | Fermented Milk (Study Group) | Unfermented Milk (Placebo Group)
Number analyzed (Participants) | 12 | 12
log10 CFU/g
  Week 0 | 7.88 (0.41) | 7.60 (0.63)
  Week 1 | 8.13 (0.49) | 8.10 (0.78)
  Week 2 | 9.03 (0.76) | 8.35 (0.59)
  Week 3 | 8.87 (0.88) | 8.11 (0.82)
  Week 4 | 9.43 (0.29) | 8.40 (0.52)
  Week 5 | 9.14 (0.45) | 8.27 (0.44)
  Week 6 | 8.51 (0.41) | 8.05 (0.63)
Statistical Analysis 1: Comparison: Fermented Milk (Study Group) vs Unfermented Milk (Placebo Group); Bacterial colonies were counted for study group and placebo group on week 0, 1, 2, 3, 4, 5, 6. Significant differences between both experimental groups at the same time were determined with one-way ANOVA (significance level p = 0.05); Test type: Superiority or Other; p < 0.05, ANOVA

2. Secondary Outcome: Modification of the Composition of the Intestinal Microflora: Escherichia Coli, Lactobacillus Spp., Lactobacillus Casei Shirota
Description: Fecal specimens were obtained from all 24 healthy volunteers at week 0, 1, 2, 3, 4, 5, 6.
  Bacterial colonies were cultured and counted.
Time Frame: at week 0, 1, 2, 3, 4, 5, 6
Reporting Status: Not Posted, anticipated posting 2009-03
Measure: Log Mean (Standard Deviation); unit: log10 CFU/g

3. Primary Outcome: Modification of the Composition of the Intestinal Microflora: Clostridium Perfringens
Description: Fecal specimens were obtained from all 24 healthy volunteers at week 0, 1, 2, 3, 4, 5, 6.
  Clostridium perfringens was cultured.Bacterial colonies were counted.
Time Frame: week 0, 1, 2, 3, 4, 5, 6.
Measure: Log Mean (Standard Deviation); unit: log10 CFU/g
Arm/Group | Fermented Milk (Study Group) | Unfermented Milk (Placebo Group)
Number analyzed (Participants) | 12 | 12
log10 CFU/g
  Week 0 | 7.13 (0.66) | 7.24 (0.59)
  Week 1 | 7.61 (0.61) | 7.57 (0.57)
  Week 2 | 8.04 (0.39) | 7.95 (0.31)
  Week 3 | 7.53 (0.69) | 7.78 (0.37)
  Week 4 | 7.29 (0.52) | 7.54 (0.43)
  Week 5 | 6.00 (0.72) | 6.83 (0.74)
  Week 6 | 6.57 (0.37) | 6.65 (0.63)
Statistical Analysis 1: Comparison: Fermented Milk (Study Group) vs Unfermented Milk (Placebo Group); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Arm/Group | Fermented Milk (Study Group) | Unfermented Milk (Placebo Group)
Serious Adverse Events (participants affected / at risk) | 0 | 0
Other Adverse Events (participants affected / at risk) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No